CLINICAL TRIAL: NCT03470792
Title: Effects of Microcirculation-assisted Adjustment of Blood Flow of Venoarterial Extracorporeal Membrane Oxygenation Life Support System on Prognosis
Brief Title: Effects of Microcirculation-assisted Adjustment of Blood Flow of VA-ECMO on Prognosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 201712044RINC
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Microcirculation; Extracorporeal Membrane Oxygenation
Keywords: Microcirculation, extracorporeal membrane oxygenation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microcirculation-assisted (Experimental): ECMO blood flow will be adjusted by conventional clinical conditions, hemodynamic parameters and microcirculation parameters
  Interventions: Device: Microcirculation examination
- Control (Active Comparator): ECMO blood flow will be adjusted by clinical conditions and conventional hemodynamic parameters
  Interventions: Device: Microcirculation examination

INTERVENTIONS:
Device: Microcirculation examination — Sublingual microcirculation images were recorded using an incident dark-field video microscope

SUMMARY:
One of the key factors of survival of patients with extra-corporeal membrane oxygenation (ECMO) life support system is whether the blood flow supplied by ECMO can meet the need of perfusion of each organ. In our previous study, we found that microcirculaton parameters within 12h after placement of venoarterial ECMO (VA-ECMO) were lower in the 28-day non-survivors than those in the survivors. Moreover, in our ongoing observational clinical trial, we found that adjustment of ECMO blood flow could improve microcirculatory dysfunction in some patients. We hypothesize that if we can find out the patients with poor microcirculation and use the microcirculation parameters to assist the adjustment of ECMO blood flow and related treatments, we might improve the survival of these patients. In this clinical trial, the patients will receive microcirculation examination within 18h after placement of ECMO. The patients were randomly divided into control and microcirculation-assisted groups. The microcirculation parameters in patients of the microcirculation-assisted group will be given to the ECMO team, and the ECMO blood flow and relative treatments will be adjusted according to macrocirculation parameters, clinical condition, and microcirculation parameters. In the patients of the control group, the ECMO blood flow and related treatments will be adjusted according to macrocirculation parameters and clinical condition. The microcirculation will be measured twice after T1, and the ECMO and related treatments will be adjusted as previous description. The microcirculation will be measured at 72h after placement of VA-ECMO. The ECMO setting, intake-output balance, dose of inotropic and vasopressors, and prognosis will be recorded. The difference will be compared between the two groups.

DETAILED DESCRIPTION:
For severe cardiac and respiratory failure patients, extra-corporeal membrane oxygenation (ECMO) life support system can help them to have time to wait for the recovery of cardiac and respiratory function or receiving advanced managements. One of the key factors of survival is whether the blood flow supplied by ECMO can meet the need of perfusion of each organ. In our previous study, we found that perfused small vessel density and proportion of perfused small vessel within 18h after placement of venoarterial ECMO (VA-ECMO) were lower in the 28-day non-survivors than those in the survivors. In one research of goal-directed treatment of septic shock, it shows that early microcirculation improved more in the patients with mild organ failure at 24h than in the patients with severe organ failure at 24h. Moreover, in our ongoing observational clinical trial, we found that adjustment of ECMO blood flow could improve microcirculatory dysfunction in some patients. We hypothesize that if we can find out the patients with poor microcirculation and use the microcirculation parameters to assist the adjustment of ECMO blood flow and related treatments, we might improve the survival of these patients. In this clinical trial, the patients will receive microcirculation examination within 18h (T1) after placement of ECMO. The patients were randomly divided into control and microcirculation-assisted groups. The microcirculation parameters in patients of the microcirculation-assisted group will be given to the ECMO team, and the ECMO blood flow and relative treatments will be adjusted according to macrocirculation parameters, clinical condition, and microcirculation parameters. In the patients of the control group, the ECMO blood flow and related treatments will be adjusted according to macrocirculation parameters and clinical condition. The microcirculation will be measured again at 6-22h after T1 and 28-44h after T1, and the ECMO and related treatments will be adjusted as previous description. The microcirculation will be measured at 72h after placement of VA-ECMO. The ECMO setting, intake-output balance, dose of inotropic and vasopressors, and prognosis will be recorded. The difference will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with venoarterial extra-corporeal membrane oxygenation

Exclusion Criteria:

* unable to receive microcirculation within 18 hours after placement of venoarterial extra-corporeal membrane oxygenation
* non-native speakers and family

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Lactate | 24h
  The difference of lactate level between Microcirculation-assisted group and control group

SECONDARY OUTCOMES:
Lactate | 48h
  The difference of lactate level between Microcirculation-assisted group and control group
Lactate | 72h
  The difference of lactate level between Microcirculation-assisted group and control group
perfused small vessel density | 24h
  The difference of perfused small vessel density between Microcirculation-assisted group and control group
perfused small vessel density | 48h
  The difference of perfused small vessel density between Microcirculation-assisted group and control group
perfused small vessel density | 72h
  The difference of perfused small vessel density between Microcirculation-assisted group and control group
endocan level | 24h
  The difference of endocan level between Microcirculation-assisted group and control group
diamine oxidase level | 24h
  The difference of diamine oxidase level between Microcirculation-assisted group and control group
inotropic score | 24h
  The difference of inotropic score between Microcirculation-assisted group and control group

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan